CLINICAL TRIAL: NCT03164941
Title: Effect of 180 Degree Selective Laser Trabeculoplasty Location on Treatment Outcomes
Brief Title: Effect of SLT Location on Treatment Outcomes
Acronym: SLOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Enitan Sogbesan, Ophthalmologist, St. Joseph's Healthcare Hamilton
Other Study IDs: 0000000000
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Glaucoma
Keywords: selective laser trabeculoplasty; practice; treatment; intraocular pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nasal SLT: This cohort will have 180 degree SLT completed on the nasal quadrants of the trabecular meshwork.
  Interventions: Procedure: Selective Laser Trabeculoplasty
- Temporal SLT: This cohort will have 180 degree SLT completed on the temporal quadrants of the trabecular meshwork.
  Interventions: Procedure: Selective Laser Trabeculoplasty

INTERVENTIONS:
Procedure: Selective Laser Trabeculoplasty — Laser treatment for glaucoma.

SUMMARY:
Selective Laser Trabeculoplasty (SLT) is a glaucoma treatment that has been shown to effectively lower intraocular pressure by increasing aqueous outflow through macrophage recruitment. There is evidence of increased drainage in the nasal quadrants of the eye. This study aims to compare whether there is a difference in the reduction of eye pressure when SLT is performed nasally and temporally.

DETAILED DESCRIPTION:
This study aims to evaluate if there is a difference between 180 degree nasal and temporal selective laser trabeculoplasty (SLT) in treatment outcomes. It is known that there is increased aqueous collectors and veins and thus aqueous drainage in the nasal quadrants of the eye. If SLT works by the hypothesized biologic mechanism in which macrophages remodel the aqueous drainage system to increase outflow, performing SLT in an area concentrated with aqueous veins may increase outflow more. As a result, we hypothesize that nasal 180 degree SLT may have better outcomes compared to the temporal counterpart. The results of this study may help inform decisions when performing 180 degree SLT and provide insight to SLT's mechanism of action. The primary objective of this study is to determine if there is a difference in treatment efficacy between nasal and temporal 180 degree SLT by measuring differences in baseline and post-operative intraocular pressures. We hypothesize that nasal SLT will have superior outcomes compared to temporal SLT due to increased number of aqueous veins.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma, ocular hypertension, pigmentary dispersion syndrome and pseudoexfoliation syndrome
* Participant must be over 18 years of age
* IOP > 16mmHg on at least two consecutive occasions separated by one month
* Two sighted eyes with visual acuity of 20/200 or better
* Informed consent from patient

Exclusion Criteria:

* Diagnosis of secondary OAG (aside from pigmentary and pseudoexfoliation glaucoma) or narrow angle glaucoma
* Previous incisional glaucoma surgery
* Incisional glaucoma surgery scheduled within 1 year of intervention
* Corneal disease affecting visualization of anterior chamber of the eye
* Treatment or plan to treat with topical or systemic steroids
* Previous selective laser trabeculoplasty treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from the glaucoma practice at St. Joseph's Healthcare Hamilton. A baseline clinical eye examination will be completed to include or exclude the participant from the study according to the criteria below. The baseline exam will include a comprehensive questionnaire of the participant's past ocular history, relevant systemic diseases, glaucoma risk factors, and surgical history.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | 1 year
  The primary outcome in this study is the change in intraocular pressure from baseline to the 1 year follow-up visit (continuous variable). The percentage decrease in IOP from baseline will also be calculated and compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- St Joseph's Healthcare Hamilton - King Campus, Hamilton, Ontario, Canada